CLINICAL TRIAL: NCT07395804
Title: DAROlutamide DoUBlet Therapy in Daily Practice (DARO-DUB) - Real-world Evaluation of Patients With Metastatic Hormone-sensitive Prostate Cancer (mHSPC) Treated With Darolutamide Plus ADT in Germany
Brief Title: How Darolutamide Plus Hormone Therapy Works for Men With Advanced Prostate Cancer in Everyday Medical Practice in Germany
Acronym: 23146
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23146
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Metastatic Hormone-sensitive Prostate Cancer (mHSPC)
MeSH Terms: interventions — darolutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Men with mHSPC fulfilling the inclusion and exclusion criteria
  Interventions: Drug: Darolutamide plus ADT treatment

INTERVENTIONS:
Drug: Darolutamide plus ADT treatment — Darolutamide + Androgen-deprivation therapy (ADT) according to local label and treating physician

SUMMARY:
Prostate cancer is a disease where cells in the prostate gland grow out of control. When prostate cancer has spread to other parts of the body but still responds to hormone treatment, it is called metastatic hormone-sensitive prostate cancer (mHSPC).

The usual treatment for this stage of prostate cancer is hormone therapy (called androgen-deprivation therapy or ADT) combined with another medicine that blocks the effect of male hormones on cancer cells, known as an androgen-receptor pathway inhibitor. Darolutamide is a newer type of androgen-receptor inhibitor.

The main goal of this study is to find out how well a combination of two treatments-darolutamide and hormone therapy (also called androgen-deprivation therapy or ADT)-works for men in Germany who have advanced prostate cancer that has spread to other parts of the body and still responds to hormone treatment. The study will look at how many men have very low or undetectable levels of a protein called prostate-specific antigen (PSA) in their blood after 12 months of treatment. PSA is a marker that doctors use to check how active prostate cancer is.

The study will also look at how long men live after starting this treatment, and will collect information about their health, the type of prostate cancer they have, and any other medicines they are taking. The study will last for 5 years. At the start of the study, the study doctor will collect information about each patient's background, such as age, other health problems, and details about their prostate cancer. This information will be taken from the patient's medical records if available. If some information is missing, the doctor may ask the patient directly.

Other information will be collected as the study goes on. This includes details about the patient's treatment, how they are doing during their regular medical visits, and any changes in their health. These check-ups and data collection will happen as part of the patient's usual care, including at the beginning of treatment, during treatment visits, follow-up visits, and at the end of the study observation period.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged ≥ 18 years
* Diagnosis of mHSPC with histological or cytological evidence for adenocarcinoma of prostate
* Metastatic disease by conventional or new generation imaging
* Physician decision to initiate treatment with Darolutamide plus ADT was made as per investigtor's routine treatment practice prior to enrollment in the study
* Signed informed patient consent before the start of data collection (according to the requirements of the local authorities and laws)

Exclusion Criteria:

* Darolutamide treatment started more than 30 days prior to study enrollment
* ADT treatment started more than 12 weeks before the start of treatment with Darolutamide plus ADT
* Hypersensitivity to Darolutamide or any other excipient
* Other prior systemic hormonal or anti-cancer treatment for mHSPC
* Participation in an investigational program for prostate cancer with interventions outside of routine clinical practice

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with metastatic hormone-sensitive mHSPC fulfilling the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2031-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with PSA < 0.2 ng/mL | 12 months

SECONDARY OUTCOMES:
Number of deaths or participants with end of observation | up to 60 months
Number of participants with PSA < 0.2 ng/mL | 3, 6, and 9 months
Number of participants with certain demographic characteristics | at study start
  * age
  * race
Number of participants with certain clinical characteristics | at study start
  * comorbities
  * Gleason score/ISUP
  * PSA prior therapy
  * prostate cancer volume and risk
  * type of metastatic disease
  * ECOG performance
Number of participants with certain testosterone value | at study start
Duration of Darolutamide + ADT treatment | up to 60 months
Timing of Darolutamide + ADT treatment start | up to 60 months
Kind of ADT treatment | up to 60 months
Number of participants who change ADT treatment | up to 60 months
Number of participants who change dosage of Darolutamide treatment | up to 60 months
Number of participants with certain reasons for Darolutamide plus ADT treatment discontinuation | up to 60 months
Number of participants with certain subsequent anti-cancer therapies | up to 60 months
Number of participants with treatment-emergent adverse events | from start of treatment up to 60 months
Number of participants with certain concomitant medication at study start and changes during treatment with Darolutamide plus ADT | up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Multiple Locations, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access. As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.